CLINICAL TRIAL: NCT00764764
Title: Shoulder Impingement: A By-Product of Cervical Spine Dysfunction?
Brief Title: Study of the Effect of Neck Treatment on Shoulder Impingement
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: CAMC Health System (Other)
Responsible Party: Clark Vaughan, CAMC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-01-2014
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2009-07

CONDITIONS: Shoulder Impingement; Shoulder Pain; Rotator Cuff Tendinitis; Cervical Degenerative Joint Disease
Keywords: shoulder pain; rotator cuff; impingement; cervical referred pain; neural tension
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Group I - Shoulder treatment only
  Interventions: Procedure: shoulder treatment
- II (Experimental): Cervical and shoulder treatment
  Interventions: Procedure: Shoulder AND cervical treatment

INTERVENTIONS:
Procedure: shoulder treatment — shoulder exercise, joint mobilization, home program, posture
  Arms: I
Procedure: Shoulder AND cervical treatment — Cervical and shoulder joint mobilization, exercise, posture, and home program
  Arms: II

SUMMARY:
The purpose of this pilot study is to conduct research to determine the most effective physical therapy treatment for a condition called shoulder impingement. This condition occurs when tissue in the shoulder is caught between the humerus (arm bone) and the scapula (shoulder blade). This causes pain when one tries to reach overhead or behind the back.

Two treatment methods will be used in the study. The first method uses the traditional treatments of hands-on shoulder stretching, shoulder exercise, posture, and education. The second method will use the traditional methods of shoulder treatment in addition to treatment of the cervical spine.

It is hypothesized that a group of patients between 40 and 70 years of age with signs and symptoms of shoulder impingement who receive physical therapy to the cervical spine and shoulder will report a higher level of functioning, will report less pain, and will gain more range of motion than a group of patients receiving physical therapy solely to the shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. the complaint of pain in either the anterior, lateral, or posterior aspect of the upper arm in an area extending from the acromion to the deltoid tubercle or to a point equally distal on the humerus.
2. production or increase in pain in any of the area(s) above with one of the following:

   1. active shoulder flexion or scaption (elevation in the scapular plane)
   2. impingement sign as described by Neer (1983)
   3. Hawkins-Kennedy impingement test (1980)
   4. resisted supraspinatus, shoulder internal or external strength testing
3. patient is between 40 and 70 years of age

Exclusion Criteria:

1. Any previous history of surgery or fracture in the cervical spine, upper thoracic spine, humerus, scapula, or clavicle
2. Any previous or current history of psychiatric or psychological treatment
3. Any medical condition that predisposes patients to shoulder pain such as past or current history of diabetes mellitus, fibromyalgia, adhesive capsulitis, rheumatoid arthritis, shoulder osteoarthritis, osteoporosis, ankylosing spondylitis, vertebrobasilar artery insufficiency, pregnancy, or shoulder instability
4. Any prolonged exposure to blood thinners or steroids
5. Constant lateral humeral pain that does not alter with movement, time of day, or position for the last 60 days
6. Subjects with an active worker's compensation claim related to the cervical spine, shoulder, or upper thoracic spine, or subjects with any impending or current litigation related to the same areas
7. A score of 11 or higher in the sensory plus affective dimensions of pain with the short-form of the McGill Pain Questionnaire
8. Any injections in the shoulder, cervical spine or upper thoracic spines in the last 6 months
9. Pain in the posterior shoulder, mid- and lower cervical spine, or upper thoracic spine that the patient wants treated
10. Onset of symptoms associated with trauma or trauma to the neck/shoulder area in the last 60 days

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Active Shoulder Scaption range of motion | 3 weeks, 6 weeks

SECONDARY OUTCOMES:
DASH Functional Questionaire | 3 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clark K Vaughan, MHSc, PT, Principal Investigator — CAMC Health System
Locations (1):
- Charleston Area Medical Center Physical Therapy and Sports Medicine, Charleston, West Virginia, United States